CLINICAL TRIAL: NCT01127568
Title: A Novel Treatment For Chronic Posttraumatic Stress Disorder (PTSD) Using Post-Reactivation Propranolol
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Douglas Mental Health University Institute (Other)
Collaborators: Massachusetts General Hospital (Other); Harvard University (Other); McGill University (Other); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Dr. Alain Brunet, Ph.D., Department of Psychiatry, Psychosocial Research Division, Douglas Mental Health University Institute, McGill University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05/25; DoD, Award #: W81XWH-08-2-0126 (Other Grant/Funding Number: U.S. Department of Defense, Award #: W81XWH-08-2-0126)
Record Dates: First submitted 2010-04-13; First posted 2010-05-21 (Estimated); Last update posted 2010-05-21 (Estimated); Status verified 2010-02

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Post-Traumatic Stress Disorders; Posttraumatic Stress Disorders; PTSD; Stress Disorder, Post Traumatic; Stress Disorders, Posttraumatic; Chronic Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propranolol (Experimental): Propranolol is a beta-blocker (blocking beta- adrenergic receptors) that reduces sympathetic activity. It is a well-known drug typically prescribed to individuals suffering from hypertension, tachycardia, cardiac arrhythmia, tremors, thyroid disease, or migraine.
  Interventions: Drug: Propranolol is available in generic form as the Wyeth product under the trade name Inderal.
- Placebo (Placebo Comparator): The placebo is an inactive capsule that will have no medication effect, but looks exactly like the medication.
  Interventions: Drug: Propranolol is available in generic form as the Wyeth product under the trade name Inderal.

INTERVENTIONS:
Drug: Propranolol is available in generic form as the Wyeth product under the trade name Inderal. — The study medication will consist of a dose of 2/3 mg/Kg of short-acting propranolol or placebo, followed 2 hours later by a dose of 1 mg/Kg of long-acting or placebo. The medication will be prescribed by the clinic's physician after medical check-up. A nurse will monitor blood pressure. According to, 40 mg of short-acting propranolol dose should produce a peak blood level of approximately 25 ng/ml at 2 hours, which the additional 60 mg long-acting propranolol should further increase by no more than 5ng. The decay of the blood level induced by the 40 mg short-acting dose after its 2-hour peak will outstrip the further rise induced by the 60 mg long-acting proposal dose, so that blood levels will not rise above this peak 30 ng/ml, which is within the therapeutic clinical range. If the participant tolerates the combination dose without any difficulty, during subsequent sessions, both the short- and long-acting doses will be given together immediately after memory reactivation.

SUMMARY:
Objective: To use propranolol to treat established chronic post traumatic stress disorder (PTSD) by reducing reconsolidation of the reactivated trauma memory.

Hypothesis: A series of treatments with propranolol, in comparison to placebo, will produce a significant reduction in PTSD symptom severity in participants with chronic PTSD.

Study Design: This is a double-blind, placebo-controlled, randomized study. Methodology: Twenty-five participants per group with chronic PTSD will be recruited. On their first visit psychodiagnostic and psychometric evaluation will take place. In addition, script-preparation for the script-driven imagery procedure will occur. Following this, the participants will return each week for a period of 6 weeks to participate in the reactivation sessions with propranolol or placebo (participants assigned to the propranolol condition will receive propranolol throughout, and participants assigned to the placebo condition will receive placebo throughout). Two weeks later, the participants will return for a follow-up of the psychodiagnostic and psychometric evaluation, as well as psychophysiological assessment using script-driven imagery procedure.

Data Analysis: A two-factor analysis of variance (ANOVA) for repeated measures will be performed on study completers. The Drug factor will have two levels: propranolol and placebo. The Time factor will have two levels: pre-treatment and post-treatment. We predict a significant Drug x Time interaction, more precisely a greater decrease in PTSD severity in the propranolol than in the placebo group. The psychophysiological data will be contrasted to a normative cutoff score for PTSD.

DETAILED DESCRIPTION:
Historical background. Recent animal research indicates that retrieval returns a consolidated memory, or some aspect(s) of it, to a labile state from which it must be restabilized in order to persist. This process is called reconsolidation, although it is not identical to consolidation. Support for reconsolidation comes from experiments in a variety of species ranging from snails to humans; in appetitive, aversive and neutral tasks; and using a broad range of approaches, including systemic or localized drug administration, gene manipulation, and interference by new learning. Memory impairments due to blocked reconsolidation can be long-lasting. Reconsolidation impairments are distinct from extinction in that they can be made to occur even when a reinforced trial is used to reactivate the memory, do not show renewal after contextual shift, can be double-dissociated from extinction, and have distinct neurochemical signatures from extinction. To date there has only been a single, published, controlled study supporting reconsolidation, and its blockade, in humans. That study involved weakening the consolidated memory of a simple motor sequence by presenting a conflicting sequence after reactivation of the memory of the original sequence.

According to a translational model of the pathogenesis of post-traumatic stress disorder (PTSD), a psychologically traumatic event overstimulates endogenous stress hormones, which in turn overly strengthen consolidation of the memory of the event, leading to an excessively powerful and persistent memory that is too easily activated, with consequent anxiety and dysfunction. Animal and human data indicate that the memory-modulating effects of stress hormones are mediated by noradrenergic activity in the amygdala and can be opposed by a β-adrenergic blocker such as propranolol. Administration of propranolol in the immediate aftermath of a psychologically traumatic event reduces the strength of its memory, as manifest in lower physiological responding during script-driven mental imagery of the event measured 3 months later, and lower self-reported PTSD symptoms measured 2 months later.

According to the above model, there exists a window of opportunity for influencing the consolidation of the traumatic event into long-term memory. Once this window has closed, the memory trace is no longer labile, and β-blockers would no longer be able to exert their anti-PTSD effect. Attempting to prevent PTSD by blocking consolidation of the traumatic memory (or some aspects of it) is subject to the formidable limitation that most cases are unlikely to receive clinical attention until long after this window of opportunity has shut. In persons who have developed PTSD, this would have happened weeks, months, or years earlier. However, if a traumatic memory undergoes reconsolidation when it is reactivated, this could re-open the window of opportunity to influence the memory pharmacologically. The post-reactivation administration of propranolol could reduce the strength of a traumatic memory by blocking reconsolidation in a manner parallel to reducing its strength immediately following its occurrence by blocking consolidation. In support of this possibility, consolidated memories for aversive tasks in animals have been shown to become sensitive to β-blockade after reactivation. Specifically, administration of propranolol following reactivation has been found to reduce inhibitory avoidance and auditory fear conditioning; the latter impairment was stable for one month. These results demonstrate in rodents that aversively conditioned memories when reactivated become sensitive to the effects of propranolol.

Previous studies supporting the proposed research. In a preliminary study, we employed a validated psychophysiological script-driven imagery technique to study 19 participants with chronic PTSD resulting from various psychologically traumatic events. Physiological responses during traumatic imagery have been shown to reliably discriminate PTSD from non-PTSD psychological trauma victims, leading to the inclusion of the PTSD criterion "physiological reactivity on exposure to internal cues that symbolize or resemble an aspect of the traumatic event" in the current Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV). Each participant described the traumatic event that caused their PTSD; this served to reactivate the traumatic memory. Immediately thereafter, the participant received either oral 40 mg short-acting propranolol followed 2 hours later by oral 60 mg long-acting propranolol (n = 9), or look-alike placebo capsules (n = 10), randomized and double-blind. Group demographic and psychometric means for the two groups were highly similar. A trained research assistant composed scripts portraying the event in the participant's own words and recorded them for playback in the laboratory.

One week later, the participant listened to an audio recording of their personal traumatic event in the psychophysiology laboratory and imagined the event as if it were happening to them again, while heart rate (HR), skin conductance (SC), and left corrugator (facial frowning muscle) electromyogram (EMG) responses were measured. Overall physiological responding during mental imagery of the traumatic event was significantly smaller in the PTSD participants who had received propranolol a week earlier compared to those who had received placebo (multivariate p = .007). Drug condition accounted for an impressive 49% of the variance in overall physiological responding. The univariate analyses indicated that HR and SC, but not EMG, responses were significantly smaller in the propranolol compared to the placebo participants. The mean HR and SC responses of the placebo participants were above the normative cut-offs for PTSD (dashed lines), whereas the mean HR and SC responses of the propranolol participants were below the normative PTSD cut-offs. The mean EMG responses of both groups fell below the normative PTSD cut-off. The observed effect sizes (in terms of Cohen's d, i.e., the difference in group means divided by the pooled standard deviation) were all in the predicted direction. By conventional standards, these effect sizes were very large for SC, large for HR, but small for EMG. The psychophysiological results of the present study along with those of the previously reported study in which propranolol was administered in the immediate aftermath of the traumatic event indicate that post-reactivation propranolol recapitulates its effects on consolidation.

Self-reported PTSD symptoms measured by the Impact of Event Scale-Revised showed a significant decline in the propranolol participants (19%), but not in the placebo participants (11%). However, the Group x Time interaction was not statistically significant, and the effect size was only moderate. Certainly the decline in self-reported PTSD symptoms in the propranolol group was less than the "decline" in physiological responses during traumatic imagery (taking the placebo group's responses as the comparison in the absence a baseline physiological measurement). However, because of their subjective nature, symptom self-reports are vulnerable to a number of potentially confounding factors, including demand effects, long-standing beliefs and expectations about oneself and one's situation, incorporating one's symptoms into one's identity, and secondary gain. All these factors may make changing self-reports more difficult than changing physiological responses, which more directly access changes in the strength of traumatic memories. It may be that anything greater than moderate improvement in PTSD symptoms is too much to ask of a single session and a single dose of propranolol.

Rationale behind the proposed research. The preliminary results described above suggest that using pharmacological consolidation blockers in conjunction with memory reactivation could have important implications for therapy. Currently cognitive behavioral therapy (CBT) which relies heavily on exposure and extinction, is the psychotherapeutic treatment of choice for anxiety disorders, including PTSD. However, its beneficial effects on PTSD -like those of drug treatment- are partial, with only one-third of patients showing lasting, clinically meaningful improvement. Modulating reconsolidation may have certain advantages over this approach. Reconsolidation blockade targets the traumatic memory directly, whereas extinction attempts to inhibit the traumatic memory through new (inhibitory) learning. There are two important drawbacks to extinction as a therapy. First, because extinction only inhibits the underlying fear memory, it will tend to spontaneously recover with the passage of time. Second, extinction is context-dependent. Thus, cognitive behavioral therapists must find ways of making extinction-based therapy context-independent and long-lasting. Otherwise, beneficial effects acquired in the office will be lost at home or over time. In contrast, reconsolidation has the theoretical advantage that impairments induced by its blockade are context-independent and long-lasting. From the practical standpoint, CBT typically requires periods of lengthy exposure to the traumatic memory or feared situation to promote extinction. In the case of reconsolidation blockade, animal research suggests that briefer exposure is more suitable.

A report of a case series of 15 patients suffering from various mental disorders who were treated with electroconvulsive therapy (ECT) claimed that when the ECT was administered during the reactivation of a memory, obsession, or hallucination, it was substantially more effective. This is roughly consistent with the possibility that psychiatric symptoms can be made to undergo reconsolidation blockade. However, the patients had a long history of psychopathology and ECT treatment, which, along with the absence of quantitative outcome measures and appropriate controls, precluded firm conclusions. Moreover, the treatment involved administration of ECT to awake patients. The practical advantage of pharmacological reconsolidation blockade over such a gross approach is obvious.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Having gone through a potentially traumatic event.

Exclusion Criteria:

* Not suffering from chronic PTSD
* Systolic blood pressure <100 mm Hg;
* Heart rate below 55 beats per minute;
* Having a medical condition that contraindicates the administration of propranolol, e.g., history of congestive heart failure, heart block, insulin-requiring diabetes, chronic bronchitis, emphysema, or asthma. With regard to asthma, because many persons who say they have had an asthma attack, especially as a child, may only have had hay fever, another allergy, or another non-asthmatic episode, a blanket exclusion criterion may be overly restrictive. Therefore, asthma attacks will only be exclusionary if they a.) occurred within the past 10 years, b.) occurred at any time in life if induced by a β-blocker, or c.) are currently being treated, regardless of the date of last occurrence. Cardiological consultation will be obtained as necessary;
* Previous adverse reaction to, or non-compliance with, a β-blocker;
* Current use of a medication that may involve potentially dangerous interactions with propranolol, including, other β-blockers, antiarrhythmics, calcium channel blockers, and potent P450 2D6 inhibitors, e.g., fluoxetine, paroxetine, miconazole, sulconazole, metoclopramide, quinidine, ticlopidine, and ritonavir. Because the protocol does not require to take large doses of propranolol on a daily basis, the decision to exclude participants will be taken by the physician on a case-by-case basis;
* Pregnancy or breast feeding. Although propranolol can be used during pregnancy we will advise women not to participate in they are or become pregnant. Women breastfeeding will also be advised not to participate because propranolol has been found in human milk. That the quantity absorbed by the breast feeding infant is inferior to 1% of the therapeutic dose (Vidal, 2008).
* Contraindicating psychiatric condition, including current psychotic, bipolar, melancholic, or substance dependence or abuse disorder; suicidality;
* Initiation of, or change in, psychotropic medication within the previous 2 months. For participants receiving stable doses of pharmacotherapy, they and their providers will be asked not to change the regimen except in clinically urgent circumstances; if this becomes necessary, a decision will be made on a case-by-case basis with regard to retaining the participant or terminating participation;
* Current participation in any psychotherapy (other than strictly supportive). Participants will be asked not to initiate psychotherapy during the course of the proposed study except in clinically urgent circumstances; if this becomes necessary, a decision will be made on a case-by-case basis with regard to retaining the participant or terminating participation;
* Inability to understand the study's procedures, risks, and side effects, or to otherwise give informed consent for participation;
* Understanding neither French nor English.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-09 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale (CAPS) for DSM-IV | Session of Week 0
  Each participant will be administered the following structured diagnostic interview instruments by a doctoral-level clinician: Clinician-Administered PTSD Scale (CAPS). The CAPS is widely regarded as the state-of-the-art structured clinical interview instrument for PTSD. It yields a categorical (present/absent) score according to DSM-IV PTSD criteria as well as severity scores for each of the 17 DSM-IV PTSD symptoms, for each of the three PTSD symptom clusters (re-experiencing, avoidance, hyperarousal) and for total PTSD.
Clinician-Administered PTSD Scale (CAPS) for DSM-IV | Session of Week 7
  Each participant will be administered the following structured diagnostic interview instruments by a doctoral-level clinician: Clinician-Administered PTSD Scale (CAPS). The CAPS is widely regarded as the state-of-the-art structured clinical interview instrument for PTSD. It yields a categorical (present/absent) score according to DSM-IV PTSD criteria as well as severity scores for each of the 17 DSM-IV PTSD symptoms, for each of the three PTSD symptom clusters (re-experiencing, avoidance, hyperarousal) and for total PTSD.
Clinician-Administered PTSD Scale (CAPS) for DSM-IV | Session of Week 26
  Each participant will be administered the following structured diagnostic interview instruments by a doctoral-level clinician: Clinician-Administered PTSD Scale (CAPS). The CAPS is widely regarded as the state-of-the-art structured clinical interview instrument for PTSD. It yields a categorical (present/absent) score according to DSM-IV PTSD criteria as well as severity scores for each of the 17 DSM-IV PTSD symptoms, for each of the three PTSD symptom clusters (re-experiencing, avoidance, hyperarousal) and for total PTSD.

SECONDARY OUTCOMES:
Mini International Neuropsychiatric Interview (MINI) | Session of Week 6
  Mini International Neuropsychiatric Interview (MINI) will evaluate pre-event history and post-event development of each Axis I mental disorder that it addresses.
Peritraumatic Distress Inventory (PDI) | Session of Week 0
  The Peritraumatic Distress Inventory (PDI) is a validated 13-item instrument that quantifies the intensity of peritraumatic emotional distress, reflecting the DSM-IV A.2 (traumatized response) PTSD criterion.
The Peritraumatic Dissociative Experiences Questionnaire | Session of Week 0
  The Peritraumatic Dissociative Experiences Questionnaire26 is a validated 10-item instrument that quantifies the intensity of dissociative reactions at the time of the traumatic event.
PTSD Check List (PCL) civilian version | Session of Week 0
  The PTSD Check List (PCL) civilian version is a scale of 17 questions that now corresponds to the DSM IV. Respondents are asked how often they have been bothered by each symptom on the past month on a 5-point severity scale.
Script-driven imagery psychophysiological measurement | Session of Week 7
  Participant will be attached to recording electrodes to measure their psychophysiological reaction while listening to the narration of a script describing their traumatic event.
PTSD Check List (PCL) civilian version | Session of Week 1
  The PTSD Check List (PCL) civilian version is a scale of 17 questions that now corresponds to the DSM IV. Respondents are asked how often they have been bothered by each symptom on the past month on a 5-point severity scale.
PTSD Check List (PCL) civilian version | Session of Week 2
  The PTSD Check List (PCL) civilian version is a scale of 17 questions that now corresponds to the DSM IV. Respondents are asked how often they have been bothered by each symptom on the past month on a 5-point severity scale.
PTSD Check List (PCL) civilian version | Session of Week 3
  The PTSD Check List (PCL) civilian version is a scale of 17 questions that now corresponds to the DSM IV. Respondents are asked how often they have been bothered by each symptom on the past month on a 5-point severity scale.
PTSD Check List (PCL) civilian version | Session of Week 4
  The PTSD Check List (PCL) civilian version is a scale of 17 questions that now corresponds to the DSM IV. Respondents are asked how often they have been bothered by each symptom on the past month on a 5-point severity scale.
PTSD Check List (PCL) civilian version | Session of Week 5
  The PTSD Check List (PCL) civilian version is a scale of 17 questions that now corresponds to the DSM IV. Respondents are asked how often they have been bothered by each symptom on the past month on a 5-point severity scale.
PTSD Check List (PCL) civilian version | Session of Week 6
  The PTSD Check List (PCL) civilian version is a scale of 17 questions that now corresponds to the DSM IV. Respondents are asked how often they have been bothered by each symptom on the past month on a 5-point severity scale.
PTSD Check List (PCL) civilian version | Session of Week 7
  The PTSD Check List (PCL) civilian version is a scale of 17 questions that now corresponds to the DSM IV. Respondents are asked how often they have been bothered by each symptom on the past month on a 5-point severity scale.
PTSD Check List (PCL) civilian version | Session of Week 26
  The PTSD Check List (PCL) civilian version is a scale of 17 questions that now corresponds to the DSM IV. Respondents are asked how often they have been bothered by each symptom on the past month on a 5-point severity scale.
Script-driven imagery psychophysiological measurement | Session of Week 26
  Participant will be attached to recording electrodes to measure their psychophysiological reaction while listening to the narration of a script describing their traumatic event.

CONTACTS AND LOCATIONS:
Overall Officials: Alain Brunet, Ph.D., Principal Investigator — Douglas Mental Health University Institute, McGill University
Locations (1):
- Douglas Mental Health University Institute, McGill University, Montreal, Quebec, Canada

REFERENCES:
- [Background] Brunet A, Orr SP, Tremblay J, Robertson K, Nader K, Pitman RK. Effect of post-retrieval propranolol on psychophysiologic responding during subsequent script-driven traumatic imagery in post-traumatic stress disorder. J Psychiatr Res. 2008 May;42(6):503-6. doi: 10.1016/j.jpsychires.2007.05.006. Epub 2007 Jun 22. PMID 17588604
- [Derived] Brunet A, Saumier D, Liu A, Streiner DL, Tremblay J, Pitman RK. Reduction of PTSD Symptoms With Pre-Reactivation Propranolol Therapy: A Randomized Controlled Trial. Am J Psychiatry. 2018 May 1;175(5):427-433. doi: 10.1176/appi.ajp.2017.17050481. Epub 2018 Jan 12. PMID 29325446
- See also: Info-trauma is an internet site with information, diagnosis and orientation for the victims of traumatic events and their loved ones. — http://www.info-trauma.org/en/home